CLINICAL TRIAL: NCT06334744
Title: Ambispective Observational Multicenter Study on the Efficacy of the Third Dose of Vaccine Anti COVID-19 in Patients Suffering From Solid Tumors Undergoing Oncological Treatment Active.
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: COVAR
Record Dates: First submitted 2024-03-26; First posted 2024-03-28 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Oncologic Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the serum neutralizing antibody titre in cancer patients undergoing active treatment against variants (VOC) before and after the third dose of BNT162b2 COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older, regardless of gender;
2. Life expectancy (estimated by the treating doctor) ≥ 6 months;
3. Histological diagnosis confirmed solid neoplasm;
4. Under active treatment
5. Previous two doses of Pfizer anti-SARS-CoV-2 vaccine received (will be considered also patients who have completed the vaccination cycle with other mRNA vaccines - Modern-)
6. All participants subscribed and signed the informed consent form first of enlistment
7. Patients with a positive history of a previous diagnosis are also enrolled laboratory confirmed COVID-19
8. ECOG 0-2

Exclusion Criteria:

1. Inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This project includes subjects affected by solid tumors undergoing active treatment and subjected to the SARS-CoV-2 vaccine belonging to MAC oncology clinics starting from the start of the vaccination campaign in fragile patients.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-01-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Determination of the change in neutralizing antibodies against SARS-CoV-2 (CLIA method) towards VOCs before the third dose of COVID-19 vaccine and 21 days after the same. | 3 weeks
  The immune response to viral variants will be evaluated by neutralization tests. In detail, previously titrated and characterized viral isolates representative of the alpha, beta, gamma and delta variants will be used. Any new variants relevant from a clinical and epidemiological point of view will subsequently be taken into consideration. A positive neutralizing titer is considered to be a titer equal to or greater than 1:10

SECONDARY OUTCOMES:
Evaluation of the kinetics of neutralizing antibodies and anti-SARS-CoV-2 IgG titer (CLIA method) up to 52 weeks after the third dose of COVID-19 vaccine | 0, 3, 26, 52 weeks
  The difference in antibody titers from time 0, at 3 and 26 weeks, up to week 52
Evaluation of the incidence of virologically confirmed cases of VOC after administration of the third dose of vaccine. | 52 weeks
  The incidence will be expressed as patients per 100 people per year.
Evaluation of the incidence of local and systemic adverse reactions (ARs), directly or indirectly linked to the vaccine, in an observation period up to 4 weeks later the third dose of vaccine. | 4 weeks
  The incidence will be expressed as patients per 100 people per year.
Evaluation of the incidence of "New onset" immune-related adverse events (IRAEs), such as immune-related pruritus, rashes, hypophysitis, hepatitis, pneumonia, diarrhoea, colitis in patients undergoing immunotherapy. | 52 weeks
  The incidence will be expressed as patients per 100 people per year.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Matteo Pavia, Pavia, PV, Italy